CLINICAL TRIAL: NCT00916383
Title: Randomized, Placebo-Controlled Study in Elderly Alzheimer's Patients on Established/Well Tolerated Dose of Aricept to Assess Skin Tolerability, Irritation, Adhesion With 3 Consecutive 7-Day Applications of 350 mg Donepezil Transdermal Patch
Brief Title: Study in Elderly Alzheimer's Patients to Assess Skin Tolerability, Irritation With 3, 7-Day Applications of DTP-System
Acronym: DTP-System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TPU-TAD-US02-0810
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2016-04

CONDITIONS: Irritation/Irritant
Keywords: Skin Irritation; Donepezil Transdermal Patch System; Elderly; Alzheimer's subjects; Skin Irritation in elderly Alzheimer's subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Upper Back (Experimental): 350 mg Donepezil Transdermal Patch (active) and placebo patch, each applied to opposite sides of the upper back.
  Interventions: Drug: 350 mg Donepezil Transdermal Patch; Drug: Placebo Patch
- Upper Arm (Experimental): 350 mg Donepezil Transdermal Patch (active) and placebo patch, each applied to opposite arms.
  Interventions: Drug: 350 mg Donepezil Transdermal Patch; Drug: Placebo Patch
- Side of Torso (Experimental): 350 mg Donepezil Transdermal Patch (active) and placebo patch, each applied to opposite sides of torso.
  Interventions: Drug: 350 mg Donepezil Transdermal Patch; Drug: Placebo Patch

INTERVENTIONS:
Drug: 350 mg Donepezil Transdermal Patch — Active and placebo patches will be applied to opposite sides for 7 days.
Drug: Placebo Patch — Active and placebo patches will be applied to opposite sides for 7 days.

SUMMARY:
This study is designed to assess skin tolerability, skin irritation, and adhesion of the 350 mg Donepezil Transdermal Patch (DTP-system), following 3, 7-day applications to 3 specific areas of the body (upper back, upper middle arm, side of torso) of elderly Alzheimer's patients. The total application time for the DTP-system is 21 days.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled study designed to evaluate skin irritation, skin tolerability, and adhesion of the 350 mg DTP-system following 3 consecutive 7-day applications to 3 specific areas of the body (upper back, upper arm, side of torso) of elderly Alzheimer's patients. The total exposure time for the DTP-system is 21 days.

All patients receive 1 Donepezil Transdermal Patch (DTP-system) and 1 placebo patch, each applied to opposite sides of the body (e.g., placebo patch to the left side of the upper back, and DTP-system to the right side of the upper back). Patients are randomized to receive the active patch to either the left or the right side of the body according to 1 of 6 treatment sequences listed below. The treatment sequence is repeated for the opposite side of the body for a total of 12 treatment sequences (4 patients in each treatment sequence). The patches are applied to one of 3 body locations for 7 days, for a total exposure period of 21 days, according to one of the following sequences:

1. Upper Back, Upper Arm, Side of Torso (Right)
2. Upper Arm, Side of Torso, Upper Back (Right)
3. Side of Torso, Upper Back, Upper Arm (Right)
4. Upper Back, Side of Torso, Upper Arm (Right)
5. Upper Arm, Upper Back, Side of Torso (Right)
6. Side of Torso, Upper Arm, Upper Back (Right)
7. Upper Back, Upper Arm, Side of Torso (Left)
8. Upper Arm, Side of Torso, Upper Back (Left)
9. Side of Torso, Upper Back, Upper Arm (Left)
10. Upper Back, Side of Torso, Upper Arm (Left)
11. Upper Arm, Upper Back, Side of Torso (Left)
12. Side of Torso, Upper Arm, Upper Back (Left)

Patches are applied on Days 1, 8, and 15 according to the randomization schedule. Oral Aricept is taken daily through Day -1, and is re-started on Day 22 or at the time of early termination if before Day 22. Patients are seen in the clinic at Screening and on Days 1, 8, 15, 22, and at the End of Study Visit; for all other daily visits, the patients may be seen either at the clinic or in their residence, provided the assessments are completed as described in the protocol. Skin irritation is assessed immediately upon patch removal and at 1, 24, and 48 hours after removal.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 65 years of age.
* Established dose of Aricept 10 mg at least 2 months prior to enrollment.
* Established diagnosis of stable Alzheimer's disease treated with oral Aricept
* Must be willing to change from oral Aricept to DTP (and placebo patch).
* Body mass index of at least 18 and a minimum weight of at least 45 kg.
* Blood pressure (sitting) must be diastolic <95mmHg, and systolic <145, stable for at least 3 months. Patients with well-controlled hypertension (with medication) may enroll as long as 3-month stability criterion is met.
* Those with stable cardiac disease may be enrolled provided the patient has been on appropriate medication for 3 months prior to screening. Those with a pacemaker may be enrolled.
* Pulse rate between 45 - 100 bpm; respirations between 8 - 20 per minute.
* Those with thyroid disease may enroll if stable on treatment for at least 3 months prior to screening, and maintain the same dose of thyroid medication throughout the study.
* Must have a caregiver who is either living with the patient or is in daily contact with the patient, agrees to be present at all visits, provide information as required, and ensure compliance with the medication schedule.
* Free from any abnormality at Screening which may compromise the patient's ability to participate.
* Free of any dermatologic conditions, excessive hair or skin allergies and sensitivities.
* Male patients who have female partners of childbearing potential must use a condom.
* Must understand and provide written informed consent (or have a Legally Authorized Representative who is able), prior to the initiation of any protocol-specific procedures.
* Must be willing and able to abide by all study requirements and restrictions.
* Must be on stable medications for at least 30 days prior to enrollment into the study.

Exclusion Criteria:

* Use of systemic or topical antihistamines within 72 hours prior to enrollment, or systemic or topical corticosteroids within 3 weeks of study enrollment or foreseen use during the study.
* History of allergy to Donepezil hydrochloride or to piperidine derivatives, related drugs, or any of the drug excipients or other drug product components.
* Those with a recent (< 2 years) cancer (except for non-melanoma skin cancers, females with in-situ cancer of the cervix or males with localized prostate cancer requiring no treatment).
* Presence of history of a psychiatric disorder, or other seizure disorder deemed clinically significant.
* Those with a known plan for elective surgery during the study period.
* Those taking antidepressant medication.
* Abnormality (e.g., scar, tattoo) or unhealthy skin (e.g., burns, wounds) at the application site; or an existing chronic skin disease or history of skin disease at the application site(s) within the 30 days prior to enrollment.
* Treatment with any investigational drug within 30 days prior to enrollment in the study.
* Any condition which would make the patient or caregiver, in the opinion of the investigator or designee, not suitable for the study for any reason.
* Current or pending legal charges that may affect patient or caregiver compliance.
* Treatment with medications contraindicated for use with Aricept

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Song, MS, MBA, Study Director — Teikoku Pharma USA, Inc.
Locations (7):
- United States (7):
  - Xenoscience, Inc, Phoenix, Arizona
  - Margolin Brain Institute, Fresno, California
  - Collaborative Neuroscience Network, Inc, Garden Grove, California
  - Synergy Clinical Research Center, National City, California
  - Apex Research Institute, Santa Ana, California
  - Meridien Research, Brooksville, Florida
  - Miami Jewish Home and Hospital for the Aged, Miami, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 clinical sites during May and June 2009. Patients received 1 placebo patch and 1 Donepezil Transdermal Patch, each applied to opposite sides of the body. The 7-day patches were applied to 1 of 3 consecutive body locations according to 1 of 6 treatment sequences for a total treatment period of 21 days.
Pre-assignment Details: Patients diagnosed with Alzheimer's disease who were on a stable course of oral Aricept (10 mg/day) were randomized into the study. Patients discontinued oral Aricept on Day -1 and resumed their original established dose following removal of the last patch.
Groups:
- All Participants: Patients were randomized to receive the active patch on the left or right side of the body, and the matching placebo patch on the same location on the opposite side of the body, and assigned to one of two sets (left and right of the body for placement of the active patch) of the following 6 treatment sequences. The treatment sequence was repeated for the opposite side of the body for a total of 12 treatment sequences. The 7-day patches were applied to one of 3 consecutive body locations, for a total exposure period of 21 days.
  1. Upper Back, Upper Arm, Side of Torso
  2. Upper Arm, Side of Torso, Upper Back
  3. Side of Torso, Upper Back, Upper Arm
  4. Upper Back, Side of Torso, Upper Arm
  5. Upper Arm, Upper Back, Side of Torso
  6. Side of Torso, Upper Arm, Upper Back
  Skin irritation scoring was obtained immediately upon removal of the patch and at 1, 24, and 48 hours after removal.
Period: Overall Study
Arm/Group | All Participants
Started | 49
Completed | 46
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All patients received the same study treatment, consisting of 1 placebo patch and 1 Donepezil Transdermal Patch, and all patches were applied to the same body locations according to 1 of 6 treatment sequences. The active patch was applied to either the right or the left side of the body according to the randomization schedule. The treatment sequence was repeated for the opposite side of the body for a total of 12 treatment sequences. The 7-day patches were applied to one of 3 body locations (upper arm, upper back, side of torso) for a total treatment period of 21 days.
Arm/Group | All Participants
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: Years]
  All Participants | 79.5 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Skin Irritation (Erythema and Edema)
Description: Erythema and edema were used to determine skin irritation using a modified Draize scale. Score 0 = no erythema/edema; Score 1 = very slight erythema/edema; Score 2 = well-defined erythema/slight edema; Score 3 = moderate to severe erythema/edema; Score 4 = severe erythema/edema.
Time Frame: Immediately after patch removal
Population: All patients who received patches are included in the analysis. Note: The represented data are based on N = 48 for patients who received the placebo patch and the DTP-system on the Upper Back, N = 46 for patients who received the placebo patch on the side of torso, and N = 47 for patients who received the DTP-system on the side of torso.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Upper Back: DTP-system and placebo patch applied to opposite sides of the upper back.
- Upper Arm: DTP-system and placebo patch applied to the upper part of opposite arms.
- Side of Torso: DTP-system and placebo patch applied to opposite sides of torso.
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 48 | 48 | 47
units on a scale
  Erythema, Placebo | 0.9 (0.85) | 0.7 (0.76) | 1.1 (0.89)
  Erythema, DTP-System | 1.0 (0.75) | 0.8 (0.75) | 1.0 (0.85)
  Edema, Placebo | 0.6 (0.82) | 0.6 (0.68) | 0.7 (0.71)
  Edema, DTP-System | 0.6 (0.76) | 0.5 (0.68) | 0.7 (0.73)

2. Primary Outcome: Skin Irritation (Erythema)
Description: Erythema was used to determine skin irritation using a modified Draize scale. Score 0 = no erythema; Score 1 = very slight erythema; Score 2 = well-defined erythema; Score 3 = moderate to severe erythema; Score 4 = severe erythema.
Time Frame: 1, 24, and 48 hours after patch removal (Days 8-10; Days 15-17; Days 22-24)
Population: All patients who received patches are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 49 | 48 | 47
units on a scale
  1 hour after patch removal, Placebo | 0.8 (0.88) | 0.6 (0.65) | 0.8 (0.82)
  1 hour after patch removal, DTP-system | 0.9 (0.73) | 0.6 (0.64) | 0.7 (0.74)
  24 hours after patch removal, Placebo | 0.6 (0.80) | 0.3 (0.52) | 0.7 (0.71)
  24 hours after patch removal, DTP-system | 0.4 (0.62) | 0.4 (0.57) | 0.4 (0.62)
  48 hours after patch removal, Placebo | 0.3 (0.54) | 0.2 (0.46) | 0.4 (0.65)
  48 hours after patch removal, DTP-system | 0.2 (0.43) | 0.2 (0.43) | 0.3 (0.59)

3. Primary Outcome: Skin Irritation (Edema)
Description: Edema was used to determine skin irritation using a modified Draize scale. Score 0 = no edema; Score 1 = very slight edema; Score 2 = slight edema; Score 3 = moderate to severe edema; Score 4 = severe edema.
Time Frame: 1, 24, and 48 hours after patch removal (Days 8-10; Days 15-17; Days 22-24)
Population: All patients who received patches are included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 49 | 48 | 47
units on a scale
  1 hour after patch removal, Placebo | 0.6 (0.76) | 0.6 (0.68) | 0.6 (0.71)
  1 hour after patch removal, DTP-system | 0.6 (0.73) | 0.4 (0.57) | 0.6 (0.71)
  24 hours after patch removal, Placebo | 0.1 (0.41) | 0.2 (0.38) | 0.2 (0.47)
  24 hours after patch removal, DTP-system | 0.1 (0.33) | 0.1 (0.34) | 0.1 (0.40)
  48 hours after patch removal, Placebo | 0.0 (0.14) | 0.0 (0.15) | 0.1 (0.25)
  48 hours after patch removal, DTP-system | 0.0 (0.14) | 0.0 (0.15) | 0.0 (0.29)

4. Primary Outcome: Skin Irritation (Papules and Vesicles)
Description: Papules and vesicles were assessed according to the following scoring criteria: Score 0 = no evidence of papules or vesicles; Score 1 = few papules or vesicles (< 10) observed on the skin site; Score 2 = more papules or vesicles (≥ 10) observed on < 50 % of skin site, diffuse or few clusters; Score 3 = many papules or vesicles observed on ≥ 50% of skin site, diffuse or few clusters; Score 4 = many papules or vesicles observed on > 50% of skin site, with multiple (> 3) clusters.
Time Frame: Immediately after patch removal
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 48 | 48 | 47
participants
  Placebo, Score >1 | 9 | 5 | 5
  DTP-System, Score >1 | 7 | 2 | 2
  Placebo, Score >2 | 2 | 1 | 1
  DTP-System, Score >2 | 1 | 0 | 0

5. Primary Outcome: Skin Irritation (Papules and Vesicles)
Description: as for outcome 4
Time Frame: 1, 24, and 48 hours after patch removal (Days 8-10; Days 15-17; Days 22-24)
Population: All patients who received patches are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 49 | 48 | 47
participants
  1 hour after patch removal, Placebo, Score >1 | 9 | 6 | 5
  1 hour after patch removal, DTP-System, Score >1 | 7 | 2 | 2
  1 hour after patch removal, Placebo, Score >2 | 2 | 1 | 1
  1 hour after patch removal, DTP-System, Score >2 | 1 | 0 | 0
  24 hours after patch removal, Placebo, Score >1 | 5 | 4 | 4
  24 hours after patch removal, DTP-System, Score >1 | 5 | 2 | 2
  24 hours after patch removal, Placebo, Score >2 | 2 | 1 | 1
  24 hours after patch removal, DTP-System, Score >2 | 0 | 0 | 0
  48 hours after patch removal, Placebo, Score >1 | 5 | 2 | 3
  48 hours after patch removal, DTP-System, Score >1 | 5 | 1 | 1
  48 hours after patch removal, Placebo, Score >2 | 2 | 1 | 1
  48 hours after patch removal, DTP-System, Score >2 | 0 | 0 | 0

6. Primary Outcome: Skin Irritation (Other Skin Effects)
Description: Other skin effects were assessed according to the following scoring criteria: Score 0 = no other effects observed; Score 1 = slight glazed appearance; Score 2 = marked glazing; Score 3 = glazing with peeling and cracking; Score 4 = glazing with fissures; Score 5 = film of dried serous exudate covering all or part of the patch site; Score 6 = small petechial erosions and/or scabs.
Time Frame: Immediately after patch removal
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 48 | 48 | 47
participants
  Placebo, Score ≥1 | 10 | 9 | 8
  DTP-System, Score ≥1 | 8 | 7 | 8
  Placebo, Score =6 | 2 | 6 | 0
  DTP-System, Score =6 | 2 | 4 | 2

7. Primary Outcome: Skin Irritation (Other Skin Effects)
Description: as for outcome 6
Time Frame: 1, 24, and 48 hours after patch removal (Days 8-10; Days 15-17; Days 22-24)
Population: All patients who received patches are included in the analysis.
Measure: Number; unit: participants
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 49 | 48 | 47
participants
  1 hour after patch removal, Placebo, Score ≥1 | 10 | 9 | 8
  1 hour after patch removal, DTP-System, Score ≥1 | 9 | 7 | 8
  1 hour after patch removal, Placebo, Score =6 | 2 | 6 | 0
  1 hour after patch removal, DTP-System, Score =6 | 3 | 4 | 2
  24 hours after patch removal, Placebo, Score ≥1 | 3 | 7 | 3
  24 hours after patch removal, DTP-System, Score ≥1 | 3 | 6 | 3
  24 hours after patch removal, Placebo, Score =6 | 2 | 5 | 1
  24 hours after patch removal, DTP-System, Score =6 | 2 | 3 | 2
  48 hours after patch removal, Placebo, Score ≥1 | 2 | 6 | 1
  48 hours after patch removal, DTP-System, Score ≥1 | 2 | 5 | 2
  48 hours after patch removal, Placebo, Score =6 | 2 | 5 | 1
  48 hours after patch removal, DTP-System, Score =6 | 2 | 3 | 2

8. Secondary Outcome: Safety, Tolerability, and Adhesion
Description: See Adverse Event section for Safety assessment. Adhesion was assessed according to the following scoring criteria: Score 0 = approximately > 90% adhered (essentially no lift off the skin); Score 1 = approximately 75% to < 90% adhered (some edges only lifting off the skin); Score 2 = approximately 50% to < 75% adhered (less than half of the system lifting off the skin); Score of 3 = approximately < 50% adhered but not detached (more than half of the system lifting off the skin without falling off); Score of 4 = Patch-system detached (patch /overlay completely off the skin).
Time Frame: Safety was assessed throughout the study. Adhesion was assessed daily and immediately prior to patch removal on Days 8, 15, and 22.
Population: Percent of Patients with Adhesion Scores <2 by Application Day
Measure: Number; unit: percentage of patients with scores <2
Arm/Group | Upper Back | Upper Arm | Side of Torso
Number analyzed (Participants) | 49 | 48 | 48
percentage of patients with scores <2
  Placebo - Worst adhesion score over 7 days | 89.6 | 93.8 | 93.8
  DTP system - Worst adhesion score over 7 days | 83.4 | 89.3 | 85.4
  Placebo - Day 1 | 97.9 | 100 | 100
  DTP system - Day 1 | 95.8 | 97.9 | 100
  Placebo - Day 2 | 100 | 100 | 100
  DTP system - Day 2 | 97.8 | 97.8 | 97.9
  Placebo - Day 3 | 100 | 97.9 | 100
  DTP system - Day 3 | 95.7 | 100 | 95.8
  Placebo - Day 4 | 100 | 95.8 | 100
  DTP system - Day 4 | 95.6 | 97.7 | 97.8
  Placebo - Day 5 | 97.9 | 100 | 100
  DTP system - Day 5 | 93.2 | 100 | 93.3
  Placebo - Day 6 | 93.5 | 97.8 | 97.9
  DTP system - Day 6 | 95.4 | 95.4 | 95.5
  Placebo - Day 7 | 91.3 | 97.8 | 95.8
  DTP system - Day 7 | 93.1 | 97.6 | 93.0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time the patient signed the Informed Consent Form until study discharge (Day 24) (3 days after removal of the last patch).
Description: All patients who received study drug were included in the safety summaries. Adverse events (AEs) collected prior to the patient receiving drug were considered baseline signs or symptoms. Any baseline sign or symptom that worsened during the course of the study was considered a treatment-emergent AE.
Groups:
- Systemic Events: All enrolled patients
- DTP-system; Placebo Patch: Localized events
Arm/Group | Systemic Events | DTP-system | Placebo Patch
Serious Adverse Events (participants affected / at risk) | 1/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 3/49 | 14/49 | 15/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Systemic Events (N=49) | DTP-system (N=49) | Placebo Patch (N=49)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Systemic Events (N=49) | DTP-system (N=49) | Placebo Patch (N=49)
Application site pruritus (General disorders) | 0 | 14 | 15
Confusional State (Psychiatric disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Institution Publication may be published provided that it does not disclose Confidential Information other than the study results from the Institution's study data. The proposed Institution Publication shall be submitted to sponsor for review and comment at least 30 days prior to submitting it to a third party. If sponsor requests a delay in order to file patent applications, the Institution Publication may be delayed for submission to a third party for up to 120 days after sponsor request.